CLINICAL TRIAL: NCT02459379
Title: Cardiac Implantable Electronic Device Magnetic Resonance Imaging Registry (CIED-MRI Registry)
Brief Title: Cardiac Implantable Electronic Device Magnetic Resonance Imaging Registry
Acronym: CIED-MRI
Status: Withdrawn | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: IDE G150066
Record Dates: First submitted 2015-05-21; First posted 2015-06-02 (Estimated); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Pacemaker Malfunction; Implantable Defibrillator Malfunction
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

INTERVENTIONS:
Radiation: MRI Scan — MRI will be performed for clinical reason for which no other imaging study will provide the data required on patients with pacemaker or implantable defibrillator

SUMMARY:
This is a prospective registry evaluating the safety of performing magnetic resonance (MRI) scans on patients who have cardiac implanted electronic devices (CIEDs). This includes pacemakers and implantable cardioverter defibrillators (ICDs). This is not a a new device approval or new MRI scanner approval, only for a registry of patients who need to have an MRI scan who already have an FDA approved CIED that is not currently labeled for use in conjunction with an MRI scan. This registry is very similar to the previously approved MagnaSafe Registry that is now closed to new enrollment.

DETAILED DESCRIPTION:
This Registry is an investigator initiated project designed to follow in the footsteps of the MagnaSafe Registry. MagaSafe was initiated to determine the risks of performing MRI for patients with pacemakers and Implantable Cardioverter-Defibrillators (ICDs). The latter is closed to new enrollments as of April 2014; however, there is still a need to accumulate data on these devices. There is also a significant clinical need, in that patients who are insured by CMS are currently excluded from having MRI scans if they have a pacemaker or ICD. The only option available to them is to undergo removal of their entire system, have the MRI scan, and then have a new system implanted. This is impossible for many patients who are "pacemaker dependent". It also exposes the patient to a well-known risk of complication from the removal/extraction process as well as the re-implant procedure. This must be contrasted to the negligible risk of having an MRI scan with the device in place (assuming proper precautions are taken), based on MagaSafe data as well as a large body of supporting literature.

Magnetic resonance is the imaging modality of choice for the diagnosis of many diseases of the brain, spinal cord, and musculoskeletal system. For some disease states, no acceptable alternative diagnostic imaging method is available. MRI is not only a superior imaging and diagnostic modality for many disorders, but also does not expose patients to ionizing radiation as does CT. The number of patients living with permanent pacemakers or ICDs is well into the millions (some estimates are up to 4 million in the US), and continues to increase. Likewise, the use of MRI continues to rise annually in all patient groups, however, as people advance in age, they are the most likely to need an MRI scan. As the device population is disproportionally weighted towards the older population, it is exactly this group that has the greatest need for MRI scans, yet may be denied.

As noted in the MagnaSafe information, "To provide optimal care to the increasing number of patients with an implanted cardiac device, health care professionals must have the capability to perform MR imaging with minimal risk and full knowledge of the possible complications." This registry recreates the protocol, safety monitoring and follow up in a manner very similar to other registries. The intent is to provide not only data that will hopefully continue to support the use of MRI scanning in device patients, but to allow this essential imaging technique to be available to patients without the need to expose them to 2 otherwise unnecessary procedures of removal and replacement of the implanted device.

This is a physician and institutional based registry that will start with New York University Langone Medical Center as collaboration between the Division of Cardiology (Electrophysiology Section) and the Department of Radiology (MRI imaging section). It is anticipated that additional sites may join in the registry over time, FDA permitting. The protocol is based on the widely published "Hopkins protocol" as attached to this submission. Several thousand patients have safely been scanned using this technique which emphasizes patient safety. Patients are monitored by experienced device personnel (ACLS certified) for vital signs (non-invasive blood pressure monitoring, pulse oximeter, and cardiac rhythm monitor (EKG)) while performing scans on patients with implanted devices. Scans are done at a major medical center equipped to manage any device or heart rhythm based complication should one occur. Only patients for whom no other imaging technique will provide adequate information are allowed to be scanned. The latter must be attested to by the physician who requires the information, and agreed upon by the electrophysiologist and the radiologist. IRB approval and a written investigator agreement will be required of any centers that may eventually participate in this registry.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age 18 or older
2. Permanent pacemaker or ICD (single, dual or multichamber), generator implanted AFTER 2001
3. Only non-MRI Conditionally Safe pacemakers and leads (but otherwise approved by the U.S. FDA ) will be included
4. Clinical indication for MRI imaging for which no other imaging modality will give adequate results to manage the patient
5. Device must have been implanted for 6 weeks or longer
6. Patient or patient's advocate must be able and willing to provide informed consent

Exclusion Criteria:

1. Presence of a lead without fixation (e.g. stand-alone SVC coil)
2. Presence of abandoned lead(s)
3. Presence of non-transvenous lead(s)
4. Other contra-indications to MRI scan (e.g. certain metallic implants)
5. Has an ICD, is pacemaker dependent, AND device not capable of asynchronous pacing mode
6. Battery voltage at replacement time indicator
7. Pacemaker or ICD labeled as MRI-Conditionally safe
8. Other contra-indication for MRI (e.g. morbid obesity, claustrophobia)
9. Pregnant patients
10. Systems that include lead adapters
11. Patients that have transvenous or transcutaneous temporary pacemaker
12. Leadless pacemakers
13. Other implants that are not compatible with MRI scans

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with CIED that is not labeled as MRI Conditionally Safe that require an MRI scan for their clinical care.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
Device function change relative to pre-scan function | Within 1 hour following the MRI Scan and at 3 months following the Scan
  Evaluation of the device post scan and then at 3 months post scan
Lead function change relative to pre-scan function | Within 1 hour following the MRI Scan and at 3 months following the Scan
  Evaluation of the lead system 1 hour post scan and then at 3 months post scan